CLINICAL TRIAL: NCT03918148
Title: Effects of Gliflozins on Markers of Cardiovascular Risk in Type 2 Diabetes (GIOIA): a Multicenter Pragmatic Prospective Cohort Study
Brief Title: Gliflozins and Cardiovascular Risk Factors in Type 2 Diabetes (GIOIA)
Acronym: GIOIA
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Katherine Esposito, Full Professor of Endocrinology and Metabolic Diseases, University of Campania Luigi Vanvitelli
Other Study IDs: 2193/2018
Record Dates: First submitted 2019-04-09; First posted 2019-04-17 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SGLT-2i: Type 2 diabetic patients treated with metformin and/or insulin starting therapy with a SGLT-2 inhibitor:
  dapagliflozin 10 mg, oral, once daily or canagliflozin 100 mg, oral, daily or empagliflozin 10 mg, oral, daily
  Interventions: Drug: SGLT-2i
- DPP-4i: Type 2 diabetic patients treated with metformin and/or insulin starting therapy with a DPP-4 inhibitor:
  sitagliptin 100 mg, oral once daily or vildagliptin 50 mg, oral, twice daily or saxaglitpin 5 mg, oral, once daily or linagliptin 5 mg, oral, once daily or alogliptin 25 mg, oral, once daily
  Interventions: Drug: DPP-4i

INTERVENTIONS:
Drug: SGLT-2i — Dapagliflozin or canagliflozin or empagliflozin add on to metformin ± basal insulin
  Groups: SGLT-2i
Drug: DPP-4i — Sitagliptin or vildagliptin or saxagliptin or linagliptin or alogliptin add on to metformin ± basal insulin
  Groups: DPP-4i

SUMMARY:
GIOIA represents a multicenter pragmatic prospective cohort study, aimed at evaluating the effects of SGLT2 inhibitors currently marketed (dapagliflozin, canagliflozin, empagliflozin) on markers of vascular, myocardial and renal damage, in patients with type 2 diabetes not well controlled with metformin and/or basal insulin. The changes of the interest outcomes are compared with those obtained with a comparator glucose lowering class (DPP-4inhibitors) over a follow-up of two years.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes for at least 5 years
* new use of an SGLT2-I or DPP4-I as add-on to metformin or insulin according to clinical practice
* HbA1c levels ≥ 7% and ≤ 8.5%
* eGFR ≥ 60 ml/min/1.73 m2

Exclusion Criteria:

* Type 1 diabetes or secondary diabetes resulting from specific causes
* History of neurovascular ulcers
* Previous therapy with SGLT-2i or DPP4-i in the 3 months prior to the study enrollment
* History of cancer within the last 5 years
* Pregnancy or active breast-feeding
* Serum creatinine level ≥ 1.3 mg/dl in women and ≥ 1.4 mg/dl in men
* eGFR ≤ 60 ml/min/1.73 m2

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with type 2 diabetes attending diabetes centers of the Campanian county treated with metformin and/or basal insulin who start therapy with a SGLT-2i or DPP-4i according to the clinical practice.
Sampling Method: Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Carotid intima-media thickness (CIMT) | 24 months
  Progression (increase in mean CIMT in millimeters [mm]) or regression (reduction > o = 0.020 mm on mean CIMT) after 2 years of follow-up
Myocardial stiffness indexes | 24 months
  Change from baseline in:
  Left Ventricular Ejection Fraction (LVEF) in percentage (%), Diastolic Left Ventricular Dimension (LVDs) in centimeters (cm) Interventricular Septum thickness (IVS) in cm left vetricular posterior wall thickness (PWs) in cm
Urinary albumin to creatinine ratio excretion | 24 months
  Development of microalbuminuria in normoalbuminuric patients at baseline or development of macroalbuminuria in patients with microalbuminuria at baseline; regression of microalbuminuria to normoalbuminuria or regression of macroalbuminuria to microalbuminuria

SECONDARY OUTCOMES:
Weight | 24 months
  Change in body weight in kilograms (kg) from baseline
Body mass index (BMI) | 24 months
  Change in body mass index in Kg/mq from baseline
Waist circumference (WC) | 24 months
  Change in waist circumference in cm from baseline
Blood pressure | 24 months
  Change in systolic and dyastolic blood pressure in mmHg from baseline
estimated Glomerular filtration rate (eGFR) | 24 months
  Change in estimated glomerular filtration rate in mI/min/1.73 mq from baseline

OTHER OUTCOMES:
HbA1c | 24 months
  Change in HbA1c in % from baseline
Mean amplitude glucose excursions (MAGE) | 24 months
  Change in MAGE in mmol/L from baseline
Lipid profile | 24 months
  Change in total cholesterol, tryglicerides, HDL-cholesterol, and LDL-cholesterol in mg/dL from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Esposito, Principal Investigator — University of Campania Luigi Vanvitelli; Dario Giugliano, Study Director — University of Campania Luigi Vanvitelli
Locations (1):
- Unit of Diabetes, Naples, Campania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giugliano D, Maiorino MI, Longo M, Esposito K. Are gliflozins the new statins for diabetes? Diabetes Res Clin Pract. 2019 Jul;153:191-193. doi: 10.1016/j.diabres.2019.04.014. Epub 2019 Apr 5. No abstract available. PMID 30959149
- [Background] Giugliano D, Maiorino MI, Bellastella G, Esposito K. Glycemic control in type 2 diabetes: from medication nonadherence to residual vascular risk. Endocrine. 2018 Jul;61(1):23-27. doi: 10.1007/s12020-017-1517-9. Epub 2018 Jan 10. PMID 29322300
- [Background] Esposito K, Longo M, Maiorino MI, Petrizzo M, Gicchino M, Bellastella G, Giugliano D. Metabolic effectiveness of gliflozins and gliptins in the routine clinical practice of patients with type 2 diabetes: preliminary results from GIOIA, a prospective multicentre study. Diabetes Res Clin Pract. 2019 Sep;155:107787. doi: 10.1016/j.diabres.2019.107787. Epub 2019 Jul 19. PMID 31326454
- [Background] Longo M, Scappaticcio L, Maiorino MI, De Nicola L, Bellastella G, Esposito K. Renal and metabolic effects of SGLT-2i and DPP-4i according to basal estimated glomerular filtration rate: Analysis from GIOIA, an observational prospective study. Diabetes Res Clin Pract. 2021 Aug;178:108990. doi: 10.1016/j.diabres.2021.108990. Epub 2021 Jul 29. PMID 34333059
- [Background] Longo M, Caruso P, Scappaticcio L, Maiorino MI, Bellastella G, Capuano A, Esposito K, Giugliano D. Two years with GIOIA 'Effects of gliflozins and gliptins on markers of cardiovascular damage in type 2 diabetes': A prospective, multicentre, quasi-experimental study on sodium-glucose cotransporter 2 and dipeptidyl peptidase-4 inhibitors in diabetes clinical practice. Diabetes Obes Metab. 2024 Apr;26(4):1492-1501. doi: 10.1111/dom.15451. Epub 2024 Jan 17. PMID 38234208